CLINICAL TRIAL: NCT05755360
Title: A Multicentre, Prospective, Non-Interventional, Single-Arm Study Investigating Glycaemic Control and Patient-Reported Outcomes in Type 2 Diabetes Patients, Uncontrolled on DPP4i Treatment and Who Switch to Oral Semaglutide in a Real-World Setting in Italy
Brief Title: DOORS: A Research Study to Understand How Oral Semaglutide Works in People With Type 2 Diabetes Who Change From Dipeptidyl Peptidase-4 Inhibitor (DPP4i) Treatment to Oral Semaglutide in Italy
Acronym: DOORS
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-7508; U1111-1274-4674 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with T2D: Participants will be treated with commercially available oral semaglutide according to routine clinical practice at the discretion of the treating physician.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will be treated with commercially available oral semaglutide according to routine clinical practice at the discretion of the treating physician. The decision to switch from DPP4i treatment to oral semaglutide is at the discretion of the treating physician and is clearly independent from the decision to include the participant in the study.

SUMMARY:
The purpose of the study is to look at the change in blood sugar levels in people with type 2 diabetes who change their treatment from DPP4i to oral semaglutide. Participant will get oral semaglutide as prescribed by the study doctor. The study will last for about 5-6 months. Participants will be asked to complete two questionnaires. One will be about eating behaviour and the other one will be diabetes related. Participant will complete this questionnaire during the normal scheduled visit with study doctor. Participants will be asked questions about their health and diabetes treatment and lab tests as part of their normal doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* The decision to switch from DPP4i treatment to commercially available oral semaglutide has been made by the participant/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the participant in this study
* Participant with last measurement of HbA1c >= 7.5% at informed consent and treatment initiation visit (V1) or less than or equal to (<=) 90 days before informed consent and treatment initiation visit (V1)
* Treatment naïve to insulin. An exception is short-term insulin treatment for acute illness for a total of < 14 days

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days prior to the informed consent and treatment initiation visit (V1) and throughout the duration of the study
* Participants with type-1 diabetes
* Participants who are pregnant or who become pregnant (or who plan to become pregnant) during the study period
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Age < 18 years on the informed consent and treatment initiation visit (V1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Participants who switch from DPP4i treatment to oral semaglutide and meet the eligibility criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Absolute change in glycated haemoglobin (HbA1c) (percentage [%]-point) | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured in %-point.
Absolute change in glycated haemoglobin (HbA1c) (millimoles per mole [mmol/mol]) | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured in mmol/mol.

SECONDARY OUTCOMES:
Relative change in body weight | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured in percentage (%).
Absolute change in body weight | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured in Kilograms (kg).
Absolute change in lipid parameters (total cholesterol, low density lipoprotein cholesterol [LDLc], high density lipoprotein cholesterol [HDLc], triglycerides) | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured in millimoles per liter (mmol/L).
Absolute change in waist circumference | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured in centimeters (cm).
Absolute change in blood pressure (systolic and diastolic) | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured in millimeters of mercury (mmHg).
Number of participants with HbA1c less than (<) 7% | At end of study (week 40 ± 4 weeks)
  Measured as number of participants (yes or no).
Number of participants with HbA1c <6.5% | At end of study (week 40 ± 4 weeks)
  Measured as number of participants (yes or no).
HbA1c reduction greater than or equal to (>=) 1%-point and body weight reduction of >= 5% | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured as number of participants (yes or no).
HbA1c reduction greater than or equal to (>=) 1%-point and body weight reduction of >= 3% | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured as number of participants (yes or no).
Self-reported severe hypoglycaemia during the study period | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  Measured as number of participants (yes or no).
Absolute change in dutch eating behaviour questionnaire (DEBQ) scores (points) | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  DEBQ is a 33-item self-reported questionnaire to assess three distinct eating behaviours in adults: emotional eating, external eating, and restrained eating. For all 33 items participants will provide response in terms of: never, seldom, sometimes, often, very often. Absolute change in DEBQ (total score) calculated as the absolute difference between the DEBQ scores (total score) at baseline and post baseline measurements of DEBQ scores (total score) up to and including end of study visit.
Absolute change in diabetes distress survey (DDS) scores (points) | From informed consent and treatment initiation (week 0) to end of study (week 40 ± 4 weeks)
  DDS is a self-administered 17-item scale that captures four critical dimensions of diabetes-related distress: emotional burden, regimen distress, interpersonal distress, and physician distress. Each item was scored in the range of 1 to 6: 1) not a problem; 2) a slight problem; 3) a moderate problem; 4) somewhat serious problem; 5) a serious problem; 6) a very serious problem. Participants will rate each item item indicating the degree to which each of the 17 items may have distressed or bothered them during the past month. High score indicated high distress.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (25):
- Italy (25):
  - Ospedale Pesenti Fenaroli, Alzano Lombardo
  - INRCA, Ancona
  - A.O.U. Policlinico S.Orsola, Bologna
  - Ospedale centrale L. Bohler, Bolzano
  - ASL Caserta, Caserta
  - Azienda Ospedaliera Cannizzaro, Catania
  - Azienda Sanitaria Locale Cn1, Cuneo
  - Università degli Studi Foggia, Foggia
  - Ospedale Misericordia, Grosseto
  - ASL Lecce, Lecce
  - Ospedale Generale provinciale, Macerata
  - Ospedale Pagliari, Massafra
  - ASL Avellino, Montoro
  - ASL Napoli 3 sud, Palma Campania
  - A.O.U. Maggiore della Carità, Piemonte
  - Ospedale San Jacopo, Pistoia
  - P.O. Praia a Mare, Praia a Mare
  - ASL Roma 2 - UOC Cure Primarie Distretto 4, Roma
  - Fondazione Univ. Policlinico A.Gemelli, Roma
  - ASL Al Di Alessandria - Ospedale Santo Spirito - Casale Monferrato - Cardiologia, Roma
  - A.O.U. Policlinico Giaccone, Sicilia
  - Casa di cure Triolo Zancla, Sicilia
  - Ospedale Treviglio, Treviglio
  - Ospedale S. Maria della Misericordia, Udine
  - ASST Sette Laghi, Varese

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com